CLINICAL TRIAL: NCT07057895
Title: Diagnostic Consistency of the Global Leadership Initiative on Malnutrition (GLIM) Criteria and the Patient-Generated Subjective Global Assessment (PG-SGA) for Malnutrition in Patients With Pancreatic Cancer
Brief Title: Diagnostic Consistency of GLIM and PG-SGA for Malnutrition in Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Feifei Wang, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022S00558
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Neoplasms
Keywords: GLIM criteria; PG-SGA; Pancreatic cancer; Malnutrition; Diagnostic consistency
MeSH Terms: conditions — Pancreatic Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Assessment Cohort (Experimental): A single cohort of patients with pancreatic cancer and nutritional risk (NRS 2002 ≥ 3) who underwent comprehensive nutritional assessment using both the GLIM criteria and the PG-SGA to evaluate the diagnostic consistency between the two tools. All participants in this arm receive all listed diagnostic procedures.
  Interventions: Diagnostic Test: Global Leadership Initiative on Malnutrition (GLIM) Criteria Assessment; Diagnostic Test: Patient-Generated Subjective Global Assessment (PG-SGA)

INTERVENTIONS:
Diagnostic Test: Global Leadership Initiative on Malnutrition (GLIM) Criteria Assessment — Malnutrition was diagnosed according to the GLIM consensus criteria. This required at least one phenotypic criterion (non-volitional weight loss, low BMI, or reduced muscle mass) and one etiologic criterion (reduced food intake/assimilation or inflammation/disease burden). Reduced muscle mass was assessed by bioelectrical impedance analysis (BIA). The assessment was performed once for each patient within 24 hours of hospital admission.
Diagnostic Test: Patient-Generated Subjective Global Assessment (PG-SGA) — A comprehensive nutritional assessment administered by trained clinical staff. The tool comprises patient-reported sections (weight history, food intake, symptoms, activities/function) and clinician-assessed sections (disease, metabolic demand, physical exam). For this study, a total score of ≥2 was considered indicative of malnutrition. The assessment was performed once for each patient within 24 hours of hospital admission.

SUMMARY:
This study aimed to evaluate the diagnostic consistency between the Global Leadership Initiative on Malnutrition (GLIM) criteria and the Patient-Generated Subjective Global Assessment (PG-SGA) for identifying malnutrition in patients with pancreatic malignant tumors. The goal is to determine if the GLIM criteria, a newer and more streamlined tool, shows substantial agreement with the well-established PG-SGA, thereby supporting its use in this high-risk clinical population.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly aggressive malignancy often associated with severe nutritional decline. While the Nutritional Risk Screening 2002 (NRS 2002) is used for initial screening and the Patient-Generated Subjective Global Assessment (PG-SGA) is a recognized standard for detailed nutritional assessment, the PG-SGA can be time-consuming. The Global Leadership Initiative on Malnutrition (GLIM) criteria were developed to provide a globally harmonized, two-step framework for diagnosing malnutrition. This prospective observational study was designed to compare the performance of GLIM criteria against the PG-SGA in patients with pancreatic cancer. Patients admitted to the hospital were screened with NRS 2002. Those at nutritional risk (NRS 2002 ≥ 3) were then comprehensively assessed using both PG-SGA and GLIM criteria. The study hypothesis is that the GLIM criteria and PG-SGA will demonstrate good consistency in diagnosing malnutrition in this population, validating GLIM as a practical and reliable assessment tool in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed pancreatic malignant tumor.
* Age ≥ 18 years.
* Clear cognition and ability to communicate verbally.
* Nutritional Risk Screening 2002 (NRS 2002) score ≥ 3.
* Provision of written informed consent to participate.

Exclusion Criteria:

* Presence of severe cardiac, hepatic, or renal comorbidities.
* Bedridden status precluding weight measurement.
* Contraindications to bioelectrical impedance analysis (e.g., implanted electronic devices, amputation).
* Concurrent diagnosis of other malignant tumors, particularly of the digestive system.
* Inability to cooperate with questionnaire completion or assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Consistency between GLIM Criteria and PG-SGA | Assessed once within 24 hours of hospital admission.
  The consistency in diagnosing malnutrition (yes/no) between the GLIM criteria and the PG-SGA was assessed. The agreement was quantified using Cohen's kappa coefficient (κ). A kappa value of 0.61-0.80 was interpreted as substantial agreement.

SECONDARY OUTCOMES:
Prevalence of Malnutrition according to GLIM Criteria | Assessed once within 24 hours of hospital admission.
  The percentage of patients diagnosed with malnutrition based on the GLIM criteria, which requires at least one phenotypic criterion (non-volitional weight loss, low BMI, or reduced muscle mass) and one etiologic criterion (reduced food intake/assimilation or inflammation/disease burden).
Prevalence of Malnutrition according to PG-SGA | Assessed once within 24 hours of hospital admission.
  The percentage of patients identified as malnourished based on the PG-SGA. A total score of ≥2 was considered indicative of malnutrition.
Correlation of Assessment Tools with Nutritional Indicators | Assessed at baseline (within 24 hours of admission).
  The correlation between the malnutrition diagnosis (by GLIM and PG-SGA) and traditional nutritional indicators was assessed using Pearson correlation analysis. The indicators included mid-upper arm circumference (AC), calf circumference (CC), Body Mass Index (BMI), serum albumin (Alb), and hemoglobin (Hb).

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China